CLINICAL TRIAL: NCT06252493
Title: Evaluation of PET/MR Enterography for Differentiation of Fibrotic and Inflammatory Strictures in Patients With Crohn's Disease Using a Collagen-binding Radiotracer.
Brief Title: Value of PET/MR Enterography in the Assessment of Crohn's Disease Using a Collagen-binding Radiotracer.
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Onofrio A. Catalano, MD, PhD, Associate Professor Harvard Medical School, PET/MR Translation Officer, Medical Director PET/MR at the Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital
Other Study IDs: 2019P001913
Record Dates: First submitted 2024-02-02; First posted 2024-02-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease
Keywords: PET/MR; Crohn Disease; [68Ga]CBP8-PET; Enterography; Fibrosis; Inflammatory Strictures
MeSH Terms: conditions — Crohn Disease; Fibrosis | interventions — Contrast Media; Magnetic Resonance Spectroscopy; Blood Specimen Collection; Glucagon; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood samples (10 ml per patient) which will be used to explore blood markers for fibrostenosis (either predictive or as biomarkers for fibrotic burden) using either serum proteomics analysis (extracellular matrix proteins using Nordic Biosciences or other proteomic platforms, e.g., Olink or similar) or serum exosome isolation for exo-miRNA profiling.
  * Tissue specimens obtained from intestinal (large and/or small bowel) surgical resections and/or endoscopic biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Crohn Disease: Patients with confirmed/suspected Crohn's disease scheduled for operative management/surgical intervention
  Interventions: Drug: Radiotracer Injection; Drug: Contrast Media, Magnetic Resonance; Diagnostic Test: Blood Draw; Drug: Glucagon; Diagnostic Test: Imaging; Drug: Oral contrast media application

INTERVENTIONS:
Drug: Radiotracer Injection — Injection of Gallium-68 labeled collagen binding probe 8 ([68Ga]CBP8):
  All subjects will undergo placement of an intravenous catheter (IV). The catheter will be flushed post-injection of [68Ga]CBP8 with 0.9% saline solution.
  The subjects will be positioned on the scanner table; support devices under the back and/or legs will be used as needed to enable the patient to comfortably maintain his/her position throughout the scan; Up to 15 mCi of [68Ga]CBP8 will be administered. The injected dose and the time of injection will be recorded;
  Post scan:
  The catheter will be removed. The subject will be asked to void again immediately after the scan and he/she will be counseled on the importance of continuing to drink fluids for several more hours in order to increase urine flow rate and minimize the radiation dose to the bladder wall.
Drug: Contrast Media, Magnetic Resonance — Dotarem 20ml will be injected during acquisition of contrast enhanced T1weighted fat saturated sequences, in keeping with standard of care MR enterography.
Diagnostic Test: Blood Draw — All subjects will undergo placement of an intravenous catheter (IV). Through the same catheter, 10 mL of venous blood will be collected to evaluate blood markers for fibrostenosis.
Drug: Glucagon — Glucagon will be injected into the subject's indwelling i.v. catheter (0.3-0.5 mg) before imaging acquisition; or intramuscularly (1-2 mg) prior to imaging the abdomen and pelvis. A second administration of IV glucagon (0.3-0.5mg) may take place during image acquisition.
Diagnostic Test: Imaging — MR and PET images of the abdomen and pelvis will be acquired using the Siemens 3 Tesla Biograph mMR scanner. Multiple anatomical and functional imaging sequences may be run to assess specific image quality measures in addition to those used for anatomical diagnosis. Among the sequences, patients will undergo a full set of standard of care MR enterography sequences to ensure they get at least same quality of study and of clinical information they would gain from a clinical study. Certain MR sequences scans may be repeated after varying a limited range of pulse sequence parameters to assess their effect on the image contrast, image artifacts and signal to noise ratio.
Drug: Oral contrast media application — Patients will be invited to drink as much as possible of an oral contrast solution consisting of a mixture of 1500-2000 ml of dilute barium or sorbitol (VoLumen or Breeza) and water. Breeza, and in the past VoLumen, is routine clinical practice at MGH. The solution comes already prepared in bottles, so there is no need to dilute or prepare. The investigators will just hand the bottle to the patient and will ask the patient to start drinking ~1 hour before the scan. By routine practice at MGH, the investigators give 3-4 bottles of Breeza, about 1500-2000ml.

SUMMARY:
In this study twenty-five (25) subjects with Crohn's disease scheduled for possible surgical intervention will be recruited for this study and a PET/MR scan using the collagen-binding radiotracer will be performed. The study aims to establish the performance figures of PET/MR using [68Ga]CBP8-PET for preoperative detection and differentiation of strictures with a fibrotic component in patients with Crohn's disease by using surgical and histologic findings (when available) as the standard for comparison. Furthermore, the investigators will determine the performance figures with which strictures are identified and characterized by PET/MR using [68Ga]CBP8-PET compared to each modality in isolation (PET alone or MR alone). Blood and tissue markers for fibrostenosis will be explored (either predictive or as biomarkers for fibrotic burden), using histologic and molecular testing by using surgical and histologic findings (when available) as the standard for comparison. Lastly the investigators want to determine the performance figures with which strictures are identified and characterized by PET/MR using [68Ga]CBP8-PET compared to each modality in isolation (PET alone or MR alone).

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a common disease affecting over 1.4 million Americans. IBD is generally further classified into one of two distinct pathologic entities: Crohn's disease and ulcerative colitis [1]. Inflammation spanning the wall of the bowel in Crohn's disease predisposes to intestinal stricture formation, which can lead to significant morbidity. Strictures in Crohn's disease are generally classified as inflammatory, fibrotic, or mixed. Differentiation between these categories has important clinical ramifications, as medical therapy is the preferred initial treatment for strictures with an inflammatory component, whereas fibrotic strictures frequently require endoscopic dilatation or surgical resection [3].

PET/MR imaging is a relatively novel imaging technique which has distinct potential advantages over conventional cross-sectional imaging (CT/MRI alone) and PET/CT imaging.The full potential of PET/MRI as an imaging modality remains largely untapped, in part due to limitation imposed by cost and time constraints of the exam. Recent advances in MR sequence technology, which allow for shorter scan times, and increased availability of combined PET/MR scanners will likely lead to an increased use of the modality in the future. The radiotracer to be used in this study is Gallium-68 labeled collagen binding probe 8 ([68Ga]CBP8), a synthetic collagen-binding probe that has already been investigated at the MGH in patients affected by pulmonary fibrosis. [68Ga]CBP8 selectively binds to collagen type I, the predominant extracellular protein in fibrosis. The deposition of type 1 collagen in the extracellular space is the final common pathway of chronic inflammation leading to irreversible end-organ architectural distortion, seen in various diseases states. There are several reasons why the improvement of current PET/MR capabilities would be beneficial. The most direct implication is that improved sensitivity and accuracy of preoperative evaluation of strictures could obviate the need for bowel resection in some cases. The immediate benefit would be avoiding the morbidity/mortality associated with a major abdominal surgery, and, in the long term, possibly avoiding or delaying dreaded complications such as short gut syndrome. Other secondary benefits are more difficult to tangibly quantify but include: 1) Reduced healthcare expenditure by avoiding use of novel biologic agents in such cases that they are unlikely to be beneficial and 2) Improved future research on therapeutic agents in Crohn's disease provided by earlier and more accurate detection of treatment response/non-response.

Twenty-five (25) subjects with Crohn's disease scheduled for possible surgical intervention will be recruited for this study. All subjects recruited for the study will be able to withdraw from the study at any time. The subjects will be referred by MGH Gastroenterology and the Crohn's and Colitis Center. The treating physician will approach the patient about the study and ask if he/she would be willing to be contacted by a member of the study staff. A study staff member will contact the recruited patients, either in person or over the phone. During the initial discussion, the investigator will explain the study in detail to the potential subject and assess inclusion/exclusion criteria. If a potential subject remains interested and meets eligibility criteria, then an appointment will be made for the subject to come to the Martinos Imaging Center in the Charlestown Navy Yard to provide informed consent and participate in the study.

All subjects will undergo placement of an intravenous catheter (IV). Through the same catheter, 10 mL of venous blood will be collected to evaluate blood markers for fibrostenosis. Study subjects will receive an injection of [68Ga]CBP8 followed by whole body MR-PET imaging acquired at 1 hour. The PET/MR scan using the collagen-binding radiotracer will be performed at the Martinos Center using the Siemens 3 Tesla Biograph mMR scanner. Standard of care MR enterography sequences will also be obtained to ensure that the subject gets at least the same quality of study and clinical information they would otherwise obtain as part of their routine pre-operative imaging. The images obtained will be interpreted by radiologists at MGH and a report will be made available in the patient's medical record. The imaging findings will be compared to operative findings and postoperative histological findings (when available). If, as part of their routine medical care as directed by their treating physician, subjects undergo endoscopic biopsies or surgery that result in pathology samples, leftover tissue, if any, will be sent to the study Sponsor, Takeda. This will only be leftover tissue handled with subjects' written consent by the Department of Pathology and judged by them as excess leftover tissue. This will not increase the time spent during surgery or endoscopy. This will not be tissue obtained for research purposes only. Takeda will use the leftover tissue to quantify the level of fibrosis in the collected tissues using a combination of H&E and Masson's trichrome stain followed by imaging profiling using spatial transcriptomics and/or multi-color imaging tools, such as CODEX through a CRO. Histopathological data will be used to establish the diagnostic accuracy, sensitivity and specificity of PET/MR using the collagen-binding probe. This will subsequently be compared to data obtained by using PET and MR enterography alone.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Biopsy confirmed/suspected Crohn's disease
* Ability to give written informed consent

Exclusion Criteria:

* Electrical implants such as cardiac pacemaker or perfusion pump;
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, or steel implants ferromagnetic objects such as jewelry or metal clips in clothing;
* eGFR of less than 30 mL/min/1.73 m2 within the past 90 days;
* Pregnant or breastfeeding (a negative quantitative serum hCG pregnancy test will be required for females of child-bearing age before the subject can participate);
* History of claustrophobia or any other condition considered likely to preclude the patient from lying comfortably in the MR/PET scanner for the duration of the exam;
* Research-related radiation exposure exceeds current Radiation Safety Committee guidelines (i.e. 50 mSv in the prior 12 months);
* BMI > 33 (limit of the PET/MR table);
* Co-morbid conditions known to cause fibrosis that may interfere with the results of the exam (e.g., retroperitoneal fibrosis, mesenteric panniculitis, desmoid tumor etc.)
* Determined by the investigator(s) to be clinically unsuitable for the study (e.g. based on screening visit and/or during study procedures);

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-five (25) subjects with Crohn's disease will be recruited for this study. The subjects will be patients with confirmed/suspected Crohn's disease scheduled for operative management/surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Detection Rate of Fibrotic Strictures with [68Ga]CBP8-PET PET/MRE. | From date of PET/MRE examination to date of final Histopathology result (1-2 Months)
  The primary endpoint of the study is to evaluate the performance of PET/MRE using [68Ga]CBP8- PET in detecting strictures containing a fibrotic component. This performance will also be compared with that of PET alone and MR enterography alone that will be acquired during the scan as well as to the findings noted at the time of surgical intervention and/or upon histologic analysis, when possible.

SECONDARY OUTCOMES:
Correlation of [68Ga]CBP8-Uptake with Degree of Fibrosis. | (1-2 Months)
  The relationship, if any, between the intensity of [68Ga]CBP8-PET uptake and degree of fibrosis will be assessed.
Detection Rate of Fibrotic Strictures with Multiparametric [68Ga]CBP8-PET/MRE. | (1-2 Months)
  The investigators will also investigate if MR derived biomarkers, for examples patterns of enhancement after gadolinium injection and ADC values might improve the performance of [68Ga]CBP8-PET.

CONTACTS AND LOCATIONS:
Overall Officials: Onofrio Catalano, MD, Ph.D, Principal Investigator — Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital, Harvard Medical School
Locations (1):
- Athinoula A. Martinos Center for Biomedical Imaging, Massachusetts General Hospital, Harvard Medical School, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham C, Cho JH. Inflammatory bowel disease. N Engl J Med. 2009 Nov 19;361(21):2066-78. doi: 10.1056/NEJMra0804647. No abstract available. PMID 19923578
- [Background] Lenze F, Wessling J, Bremer J, Ullerich H, Spieker T, Weckesser M, Gonschorrek S, Kannengiesser K, Rijcken E, Heidemann J, Luegering A, Schober O, Domschke W, Kucharzik T, Maaser C. Detection and differentiation of inflammatory versus fibromatous Crohn's disease strictures: prospective comparison of 18F-FDG-PET/CT, MR-enteroclysis, and transabdominal ultrasound versus endoscopic/histologic evaluation. Inflamm Bowel Dis. 2012 Dec;18(12):2252-60. doi: 10.1002/ibd.22930. Epub 2012 Feb 22. PMID 22359277
- [Background] Catalano OA, Gee MS, Nicolai E, Selvaggi F, Pellino G, Cuocolo A, Luongo A, Catalano M, Rosen BR, Gervais D, Vangel MG, Soricelli A, Salvatore M. Evaluation of Quantitative PET/MR Enterography Biomarkers for Discrimination of Inflammatory Strictures from Fibrotic Strictures in Crohn Disease. Radiology. 2016 Mar;278(3):792-800. doi: 10.1148/radiol.2015150566. Epub 2015 Oct 5. PMID 26436860
- [Background] Catalano OA, Wu V, Mahmood U, Signore A, Vangel M, Soricelli A, Salvatore M, Gervais D, Rosen BR. Diagnostic performance of PET/MR in the evaluation of active inflammation in Crohn disease. Am J Nucl Med Mol Imaging. 2018 Feb 5;8(1):62-69. eCollection 2018. PMID 29531862
- [Background] Pellino G, Nicolai E, Catalano OA, Campione S, D'Armiento FP, Salvatore M, Cuocolo A, Selvaggi F. PET/MR Versus PET/CT Imaging: Impact on the Clinical Management of Small-Bowel Crohn's Disease. J Crohns Colitis. 2016 Mar;10(3):277-85. doi: 10.1093/ecco-jcc/jjv207. Epub 2015 Nov 15. PMID 26574490
- [Background] Desogere P, Tapias LF, Hariri LP, Rotile NJ, Rietz TA, Probst CK, Blasi F, Day H, Mino-Kenudson M, Weinreb P, Violette SM, Fuchs BC, Tager AM, Lanuti M, Caravan P. Type I collagen-targeted PET probe for pulmonary fibrosis detection and staging in preclinical models. Sci Transl Med. 2017 Apr 5;9(384):eaaf4696. doi: 10.1126/scitranslmed.aaf4696. PMID 28381537